CLINICAL TRIAL: NCT02195648
Title: Treatment Efficacy of Tension Type Headache After Application of Sub-occipital Muscle Inhibition Technique Associated With Interferential Electrotherapy
Brief Title: Sub-occipital Muscle Inhibition in Tension Type Headache
Acronym: TTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Raúl Pérez Llanes, Diplomado en Fisioterapia, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: tension type headache
Record Dates: First submitted 2014-07-15; First posted 2014-07-21 (Estimated); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Tension-Type Headache
Keywords: Tension-Type Headache; Physical Therapy Modalities; Musculoskeletal Manipulations; Sub-occipital muscle inhibition technique
MeSH Terms: conditions — Tension-Type Headache

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcome assessor will be blinded to group allocation. Additionally, analysis blinding will be performed to group allocation.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Suboccipital inhibition (Experimental): The intervention group will receive a session of 20 minutes (5 minutes for the patient's reception, 10 for treatment and the following 5 minutes for rest and hemodynamic stabilization), twice a week for 4 weeks. The intervention will consist of suboccipital muscle inhibition and interferential current on the occipital muscles.
  Interventions: Other: Suboccipital inhibition
- Control (No Intervention): No intervention will be done to the participants during the study. After study completion, the participants will be offered to receive the therapy.

INTERVENTIONS:
Other: Suboccipital inhibition — Experimental: Suboccipital inhibition
  The intervention group will receive a session of 20 minutes (5 minutes for the patient's reception, 10 for treatment and the following 5 minutes for rest and hemodynamic stabilization), twice a week for 4 weeks. The intervention will consist of suboccipital muscle inhibition and interferential current on the occipital muscles.
  Arms: Suboccipital inhibition

SUMMARY:
The main objective of this study is to determine the effects caused in neck movement, neck pain, headache in patients with tension type headache and cervicogenic headache after application of sub-occipital muscle inhibition technique associated with interferential electrotherapy.

DETAILED DESCRIPTION:
This study is based on the combined application of sub-occipital muscle inhibition technique associated with interferential electrotherapy improves symptoms in patients with tension type headache and cervicogenic headache.

The purposes of this study are:

* Evaluate the effectiveness of treatment based on the combined application of sub-occipital muscle inhibition technique associated with interferential electrotherapy in patients with tension type headache.
* Evaluate the effects of treatment caused in upper cervical movement.
* Evaluate the effects of treatment caused in neck pain.
* Evaluate the effects of treatment caused in headache.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with tension type headache
* In prophylactic regimen and with medical control

Exclusion Criteria:

* Patients with neurological or cognitive impairments that prevent understanding the questionnaires
* Patients diagnosed with other types of headaches
* Patients who have not signed the informed consent document

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-02; Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Pain | Pain will be assessed at baseline, before and after each session (twice a week for 4 weeks)
  Our primary outcome will consist of changes at each session in self-reported pain, which will be measured with a visual analogic scale (VAS).
Anxiety | STAI will be assessed at baseline and after 4 weeks.
  Anxiety will be assessed with the State-Trait Anxiety Inventory. This questionnaire is designed for the self-assessment of anxiety (Cronbach's α for this scale ranges from .83 to .92).

SECONDARY OUTCOMES:
Headache Disability | HDI will be assessed at baseline and after 4 weeks.
  The Spanish version of the Headache Disability Inventory (HDI) which has shown a strong consistency/reliability will be used to measure neck disability. The HDI consists of 25 items assessing emotional (13 items) and functional aspects (12 items) with 4 possible response options, the total score ranging from 0 to 52 points and 0 to 48 points for emotional and functional aspects, respectively, with higher scores indicating more disability.
Headache Impact Test | HIT-6 will be assessed at baseline and after 4 weeks.
  The impact of headache on daily life will be measured by the Headache Impact Test-6 (HIT-6) (Cronbach alpha 0.89; test-retest reliability ranging from 0.78 to 0.90). The HIT-6 consists of 6 items with 4 response options. The total score of HIT-6 ranging from 36 to 78 points, where a higher score indicates a greater impact of headache on the daily life of the respondent.
Range of Motion | ROM will be assessed at baseline and after 4 weeks.
  Upper cervical range of motion will be measured with the CROM-device (Performance Attainment Associates. 958 Lydia Drive, Roseville, Minnesota, USA. 55113) which has demonstrated a good intra-tester reliability for cervical extension, flexion, lateral flexion and rotation. The flexion, extension and lateral flexion ranges of motion will be measured actively with the patient sit in a straight-back chair. The subject will be instructed to move their head and neck through all cardinal planes. The range of motionwill be determined either by the patient reporting the onset of pain or firm resistance met by the evaluator. Three measurements will be done, and the average will be selected for future analysis.
Neck Disability Index | NDI will be assessed at baseline and after 4 weeks.
  Neck Dissability Index (NDI) is a modification of the Oswestry low back pain disability index, and has the most commonly used self-report measure for neck pain. It is a patient-completed, condition-specific functional status questionnaire with 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation. The tool is 5-ordinal scale from 1 (I can't) to 5 (I can), with a maximum score 50.
  The NDI has good reliability and validity in persons with mechanical neck pain.
SF-36 Health Survey | SF-36 will be assessed at baseline and after 4 weeks.
  The SF36 is a shortened version of a battery of 149 health status questions developed and tested on a population of over 22,000 patients as part of the medical outcome study.
Depression | BECK II will be assessed at baseline and after 4 weeks.
  BECK II will be used to measure the participant's depression. The Beck Depression Inventory consists of 21 items, assessing depressive symptoms on a Likert scale of 0-3, ranging from 0 = "rarely or not at all" to 3 = "most of the time or always", with overall scores ranging from 0 to a maximum of 63 points.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Meroño-Gallut, PhD, Study Director — Universidad Católica San Antonio de Murcia
Locations (1):
- Universidad Católica San Antonio de Murcia, Murcia, Guadalupe, Spain